CLINICAL TRIAL: NCT06506305
Title: A Single/Multiple Dose Escalation, Open-Labeled, Phase I Clinical Study to Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of FB1001 in Patients With Acute Optic Neuropathy
Brief Title: Clinical Study of FB1001 in Patients
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: 4B Technologies Limited (Industry)
Responsible Party: Principal Investigator, Xiaodong Sun, Director, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FB1001-03-101
Record Dates: First submitted 2024-05-21; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Optic Neuropathy; NAION - Non-Arteritic Ischemic Optic Neuropathy; APAC - Acute Primary Angle Closure; Glaucoma, Angle-Closure
MeSH Terms: conditions — Optic Nerve Diseases; Glaucoma, Angle-Closure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- SAD Cohort 1 (Experimental): Participants in this cohort will receive SAD dose 1 of FB1001
  Interventions: Drug: FB1001
- SAD Cohort 2 (Experimental): Participants in this cohort will receive SAD dose 2 of FB1001
  Interventions: Drug: FB1001
- SAD Cohort 3 (Experimental): Participants in this cohort will receive SAD dose 3 of FB1001
  Interventions: Drug: FB1001
- Experimental: SAD Cohort 4 (Experimental): Participants in this cohort will receive SAD dose 4 of FB1001
  Interventions: Drug: FB1001
- Experimental: SAD Cohort 5 (Experimental): Participants in this cohort will receive SAD dose 5 of FB1001
  Interventions: Drug: FB1001
- Experimental: MAD Cohort 1 (Experimental): Participants in this cohort will receive MAD dose 1 of FB1001
  Interventions: Drug: FB1001
- Experimental: MAD Cohort 2 (Experimental): Participants in this cohort will receive MAD dose 2 of FB1001
  Interventions: Drug: FB1001
- Experimental: MAD Cohort 3 (Experimental): Participants in this cohort will receive MAD dose 3 of FB1001
  Interventions: Drug: FB1001

INTERVENTIONS:
Drug: FB1001 — Intravitreal (IVT) injection

SUMMARY:
This study is designed for single-center, open-label, dose escalation phase I trial to evaluate the safety and tolerability of a single/multiple intravitreal injection of FB1001 in patients with APACG(Acute Primary Angle-Closure Glaucoma) or NAION(Nonarteritic Anterior Ischemic Optic Neuropathy).

DETAILED DESCRIPTION:
After acute attack of APACG or NAION, patients are going to experience progression of visual field or visual acuity defects, even after IOP or inflammation control by diverse treatments. FB1001 is a recombinant humanized monoclonal antibody that protects and repairs the optic nerve, thereby delaying the progression of glaucoma and NAION. The main purpose of this study is to evaluate the safety and tolerability of FB1001 by single/multiple intravitreal injections to Acute Optic Neuropathy Patients. Pharmacokinetic profile through blood/Aqueous will be investigated and preliminary efficacy will be explored if possible. SAD(Single Ascending Dose) will consist of a maximum of 5 cohorts and each cohort will enroll 3 to 6 eligible patients. MAD(Multiple Ascending Dose) will consist of a maximum of 3 cohorts and each cohort will enroll 8 eligible patients. For each participant, the study will last up to about 12 weeks for SAD part, and 24 weeks for MAD part.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Acute Primary Angle-Closure Glaucoma (APACG) Optic Neuropathy：

   1. Within 120 hours prior to the planned administration of the study drug, the study eye has the initial symptoms of an acute attack of primary angle closure; refer to the diagnostic criteria as attached in protocol;
   2. The symptom duration of the acute attack ≥1 day, and the experienced highest intraocular pressure (IOP) in the study eye ≥30 mmHg;
   3. After acute attack is controlled, the BCVA in the study eye is 20/40 or higher;
   4. After successful treatment of the acute attack, the IOP of the study eye <21 mmHg before dosing.
2. Patients with Acute Non-arteritic Anterior Ischemic Optic Neuropathy (NAION)

   1. Positive diagnosis of NAION with symptom onset within 14 days prior to planned dosing with FB1001, refer to the diagnostic criteria as attached in protocol;
   2. Before drug administration, the BCVA score in the study eye by ETDRS is better than or equal to 15 letters.
   3. The use of corticosteroids remains stable before and after drug administration (Dose adjust determined by investigator, if needed).
3. At least 40 years old;
4. Sufficiently clear ocular media and adequate pupil dilation to allow observation and assessment of the optic nerve and macula in the study eye;
5. Female subjects of childbearing potential, and male subjects with partners of childbearing potential, should agree to use effective contraception from the time of signing the informed consent form until 3 months after the last drug administration.

Exclusion Criteria:

1. Patients with Acute Primary Angle-Closure Glaucoma (APACG) Optic Neuropathy:

   1. History or current diagnosis of glaucoma in both eyes;
   2. History of chronic primary angle-closure glaucoma in any eye;
   3. History of secondary angle-closure glaucoma in any eye.
2. Patients with Acute Non-arteritic Anterior Ischemic Optic Neuropathy (NAION):Intraocular pressure >24 mmHg in the study eye;

   1. History of optic neuritis or uveitis in any eye;
   2. Clinical evidence of temporal arteritis;
   3. History of collagen vascular disease or other inflammatory disease, or multiple sclerosis;
   4. Currently diagnosed with NAION in both eyes.
   5. The treatment with compound papaverine-like drugs is less than 5 half-lives from the administration of the study drug.
3. The study eye has opacities of the refractive media or miosis that affect fundus examination, as judged by the investigator to be unsuitable for inclusion;
4. The equivalent sphere of the refractive error in the study eye exceeds 6.0 diopters;
5. The study eye has any ocular disease or past history that may affect vision and/or visual field other than acute angle-closure glaucoma and NAION [Vitreomacular traction syndrome, retinal detachment, Age-related macular degeneration, Retinal vein occlusion, Macular hole, Epiretinal membrane, Retinal pigment epithelial tear involving the macula, Diabetic retinopathy (except for mild non-proliferative diabetic retinopathy that does not require treatment), Optic neuritis, etc.], as judged by the investigator to be unsuitable for inclusion;
6. The study eye has previously undergone subfoveal laser coagulation, vitrectomy, macular translocation surgery, or transpupillary thermotherapy;
7. The study eye has undergone intraocular surgery (such as intraocular lens implantation, etc.) or periocular surgery within 90 days before drug administration, or eyelid surgery within 30 days before drug administration;
8. The study eye has undergone YAG laser posterior capsulotomy within 28 days before drug administration;
9. History of surgical procedure within 1 month before screening, and/or currently has unhealed wounds, ulcers, fractures, etc., and is judged by the investigator to be unsuitable for inclusion;
10. The study eye has received intraocular or peribulbar injection of corticosteroids (such as triamcinolone, etc.) within 6 months before screening;
11. Continuous use of systemic corticosteroids for more than 1 week within 90 days before drug administration (except for systemic steroid treatment for NAION before screening);
12. Any eye has received any intravitreal anti-VEGF treatment (such as bevacizumab, aflibercept, etc.) within 90 days before drug administration;
13. Any eye has a history of active ocular inflammation or infection within 30 days before drug administration;
14. Presence of infectious diseases requiring systemic treatment (oral, intramuscular, or intravenous medication) before screening;
15. Systemic application of nerve growth factor or BDNF-like treatment within 90 days before drug administration;
16. Participation in any clinical trial for the treatment of optic neuropathy within 90 days before drug administration, with the exception of dietary supplements, vitamins, or minerals;
17. Participation in any clinical trial within 60 days before drug administration;
18. History of allergic reaction to fluorescein and indocyanine green, history of allergy to therapeutic or diagnostic biological products, or allergy to the study drug or its components.
19. Currently using or likely to require systemic medication that may cause crystalline or retinal toxicity, such as deferoxamine, chloroquine/hydroxychloroquine, tamoxifen, phenothiazine, and ethambutol, etc.;
20. History of myocardial infarction, unstable angina, coronary revascularization within 6 months before screening, cerebrovascular accident history (including TIA), other thromboembolic disease history (such as thromboangiitis, pulmonary embolism, deep vein thrombosis, portal vein thrombosis, etc.), New York Heart Association (NYHA) class ≥II heart failure, severe arrhythmia;
21. Presence of systemic autoimmune diseases;
22. Presence of disseminated intravascular coagulation and significant bleeding tendency (such as hemoptysis, hematemesis, severe purpura, etc.) within 3 months before screening, or having received anticoagulant or antiplatelet treatment other than aspirin/NSAIDs within 14 days before screening; Blood PLT ≤ 100 × 10^9/L, prothrombin time and activated partial thromboplastin time ≥ 3 seconds above the normal range (based on the normal values of the clinical trial institution's laboratory); taking antiplatelet drugs or anticoagulant drugs within 1 month before screening (patients taking a daily dose of aspirin ≤ 100mg are not included in this anticoagulant requirement, for patients taking aspirin, it is allowed to adjust the dose to 100mg and below on the day before screening to proceed with screening);
23. Combined with severe liver and kidney diseases, or abnormal liver and kidney function during the screening period (ALT, AST ≥ 2.5 times the upper limit of the normal value; total bilirubin ≥ 1.5 times the upper limit of the normal value; creatinine, urea/blood urea nitrogen ≥ 1.2 times the upper limit of the normal value);
24. Poorly controlled hypertension, defined as a single measurement of systolic blood pressure >180 mmHg, or two consecutive measurements of systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg (with a time interval of ≥30 minutes between measurements);
25. Women who are already pregnant during the screening period, or are in the pregnancy or lactation period;
26. Presence of active malignant tumors or a history of malignant tumors within 5 years before the baseline visit, except for completely cured in situ cervical cancer, and completely cured and regressed non-metastatic skin squamous cell carcinoma or basal cell carcinoma;
27. History of mental illness, family history of mental illness, or emotional disorders as judged by the investigator or a psychiatrist;
28. Other situations to be excluded judged by the investigator.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
SAD phase: DLTs incidence | within 28 days after dosing
  DLTs observed during the DLT observation period
SAD phase: Incidence of Treatment-Emergent Adverse Events | Baseline to 12 weeks
  The percentages of subjects experiencing AEs will be calculated.
MAD phase: Incidence of Treatment-Emergent Adverse Events | Baseline to 24 weeks
  The percentages of subjects experiencing AEs will be calculated.

SECONDARY OUTCOMES:
AUC0-t | Baseline to end of study, SAD up to 12 weeks and MAD up to 24 weeks
  The area under the drug-time curve from 0 to time t
AUC0-∞ | Baseline to end of study, SAD up to 12 weeks and MAD up to 24 weeks
  The area under the curve at the time of 0-infinity
Cmax | Baseline to end of study, SAD up to 12 weeks and MAD up to 24 weeks
  The peak concentration
Tmax | Baseline to end of study, SAD up to 12 weeks and MAD up to 24 weeks
  The peak time
CL | Baseline to end of study, SAD up to 12 weeks and MAD up to 24 weeks
  Clearance rate
t1/2 | Baseline to end of study, SAD up to 12 weeks and MAD up to 24 weeks
  Half-life
MAD phase: Cmin,ss | Baseline to 24 weeks
  The trough concentration in steady state
MAD phase: Cavg,ss | Baseline to 24 weeks
  The average concentration in steady state
MAD phase: Rac | Baseline to 24 weeks
  Accumulation Index
Immunogenicity evaluation indicators | Baseline to end of study, SAD up to 12 weeks and MAD up to 24 weeks
  Positive rate of anti-drug antibody. (neutralizing antibody, if needed)
Preliminary biological effects and efficacy evaluation indicator 1 | Baseline to end of study, SAD up to 12 weeks and MAD up to 24 weeks
  Anatomical changes in optic nerve head by OCT compared with baseline/fellow eyes
Preliminary biological effects and efficacy evaluation indicator 2 | Baseline to end of study, SAD up to 12 weeks and MAD up to 24 weeks
  Changes in RNFL thickness by OCT with baseline/fellow eyes
Preliminary biological effects and efficacy evaluation indicator 3 | Baseline to end of study, SAD up to 12 weeks and MAD up to 24 weeks
  Changes in GCC by OCT compared with baseline/fellow eyes
Preliminary biological effects and efficacy evaluation indicator 4 | Baseline to end of study, SAD up to 12 weeks and MAD up to 24 weeks
  Changes in blood flow density of optic disc by OCTA with baseline/fellow eyes
Preliminary biological effects and efficacy evaluation indicator 5 | Baseline to end of study, SAD up to 12 weeks and MAD up to 24 weeks
  Changes in blood flow density of macula by OCTA with baseline/fellow eyes
Preliminary biological effects and efficacy evaluation indicator 6 | Baseline to end of study, SAD up to 12 weeks and MAD up to 24 weeks
  Changes in BCVA/Visual Field compared with baseline
Preliminary biological effects and efficacy evaluation indicator 7 | Baseline to end of study, SAD up to 12 weeks and MAD up to 24 weeks
  Changes in P-VEP(pattern-visual evoked potential)compared with baseline
Preliminary biological effects and efficacy evaluation indicator 8 | Baseline to end of study, SAD up to 12 weeks and MAD up to 24 weeks
  Changes in P-ERG compared with baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai Jiao Tong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
After the data is published, the IPD will be shared.